CLINICAL TRIAL: NCT01341132
Title: Evaluation of Cirrhosis and Malignant Hepatic Lesions Using Novel MR Contrast Agents
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Bayer Healthcare Pharmaceuticals, Inc./Bayer Schering Pharma (Industry); University of California, San Francisco (Other)
Responsible Party: Rizwan Aslam, San Francisco Veterans Administration Medical Center
Other Study IDs: 10-03278
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: HCC; Hepatocellular Carcinoma; MRI; Liver
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — gadolinium ethoxybenzyl DTPA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Suspected Liver Disease: 1. Alpha-feto protein > 400 ng / mL or
  2. prior ultrasound with mass suspicious for hepatic malignancy or.
  3. clinical risk of hepatocellular carcinoma or
  4. prior multi-detector CT with mass suspicious for possible hepatocellular carcinoma
  Interventions: Procedure: MRI Scan of the Liver enhanced with Eovist

INTERVENTIONS:
Procedure: MRI Scan of the Liver enhanced with Eovist — 10mL of gadoxetate disodium administered intravenously while being scanned via the MRI. Images will be attained on a 5, 10 and 20 minute delay. Expected scan time is 45 minutes total

SUMMARY:
This study aims to determine whether or not gadoxetate disodium (Eovist) enhanced magnetic resonance imaging (MRI) has a higher sensitivity for detecting hepatocellular carcinoma (Liver Cancer) comparison to multi-detector computed tomography (CT).

ELIGIBILITY:
Inclusion Criteria:

* Alpha-feto protein > 400 ng / mL or
* prior ultrasound with mass suspicious for hepatic malignancy or.
* clinical risk of hepatocellular carcinoma or
* prior multi-detector CT with mass suspicious for possible hepatocellular carcinoma

Exclusion Criteria:

* Glomerulo-filtration rate < 50 mL/ min/1.73 m2 based on a creatinine measurement within three months of the MR study
* Previous diagnosis of hepatic malignancy
* Any conditions that would discount the ability to have an MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 75 patients of the San Francisco VA Medical Center with suspected HCC identified on contrast-enhanced multi-detector CT, or on ultrasound and referred to contrast-enhanced multi-detector CT.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rizwan Aslam, MD, Principal Investigator — San Francisco VA Medical Center
Locations (1):
- San Francisco VA Medical Center, San Francisco, California, United States